CLINICAL TRIAL: NCT05487248
Title: A Study of On-treatment ctDNA Changes in Chemo-refractory Colorectal Cancer Patients
Acronym: COPERNIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IJB-COPERNIC-ODN-012
Record Dates: First submitted 2022-05-27; First posted 2022-08-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Unresectable Locally Advanced Colorectal Cancer; Metastatic Colorectal Cancer; Candidate for Third-line or Subsequent Lines of Therapy
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unresectable locally advanced or metastatic colorectal cancer patients (Experimental): ● Samples collection:
  Blood samples 2 x 9 ml at day 1 2 x 9ml at day 15
  Plasma samples 2 x 9 ml at day 1 4 x 9 ml at day 29 4 x 9 ml at week 8 or 12 and every 8 or 12 weeks thereafter (+/- 7 days) until evidence of progressive disease by RECIST 1.1 (according to local assessment)
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — For subjects receiving treatments with a 2- or 4-weekly schedule, samples for ctDNA testing will be collected at the following timepoints:
  Blood :
  * Before treatment start (day 1)
  * 2 weeks after treatment start (day 15)
  Plasma :
  * Before the treatment start (day 1)
  * 4 weeks after treatment start (day 29)
  * 8 or 12 weeks after treatment start and every 8 or 12 weeks thereafter (i.e. at the same time of each imaging tumour assessment) until evidence of progressive disease by RECIST 1.1
  For subjects receiving treatments with a 3-weekly schedule, samples for ctDNA testing will be collected at the following timepoints:
  Blood :
  * Before treatment start (day 1)
  * 3 weeks after treatment start (day 22)
  Plasma :
  * Before treatment start (day 1)
  * 6 weeks after treatment start (day 43)
  * 8 or 12 weeks after treatment start and every 8 or 12 weeks thereafter (i.e. at the same time of each imaging tumour assessment) until evidence of progressive disease by RECIST 1.1

SUMMARY:
COPERNIC is an international, multicentre, single-arm study. Chemo-refractory mCRC subjects who meet all eligibility criteria will be treated with standard systemic chemotherapy (the decision about the treatment regimen being made by the treating physician) and undergo tumour assessment by standard imaging (either CT scan or MRI scan) at baseline and every 8 or 12 weeks until evidence of tumour progression. Response to treatment will be assessed by the local investigators according to the RECIST criteria version 1.1. Blinded, independent central review of the imaging scan will be carried out, this having no impact on treatment decisions thatwhich will remain the prerogative of the treating physician.

Serial blood samples from study subjects will be collected at pre-defined time points for ctDNA testing. Also, archived tumour tissue from each subject will be collected. Prospective and retrospective ctDNA analyses on blood samples will be carried out, and dynamics of ctDNA will be correlated with treatment outcomes prognosis.

DETAILED DESCRIPTION:
COPERNIC is an international, multicentre, single-arm study. Chemo-refractory mCRC subjects who meet all eligibility criteria will be treated with standard systemic chemotherapy (the decision about the treatment regimen being made by the treating physician) and undergo tumour assessment by standard imaging (either CT scan or MRI scan) at baseline and every 8 or 12 weeks until evidence of tumour progression. Response to treatment will be assessed by the local investigators according to the RECIST criteria version 1.1. Blinded, independent central review of the imaging scan will be carried out, this having no impact on treatment decisions which will remain the prerogative of the treating physician.

Serial blood samples from study subjects will be collected at pre-defined time points for ctDNA testing. Also, archived tumour tissue from each subject will be collected. Prospective and retrospective ctDNA analyses on blood samples will be carried out, and dynamics of ctDNA will be correlated with prognosis.

Two ctDNA assays will be used in this study:

* FoundationOne Liquid CDx (F1LCDx) for comprehensive genomic profile (CGP) assessment
* F1Monitor for monitoring purpose

For subjects receiving treatments with a 2- or 4-weekly schedule, blood and plasma samples for ctDNA testing will be collected at the following timepoints:

Blood :

* Before treatment start (day 1)
* 2 weeks after treatment start (day 15)

Plasma :

* Before the treatment start (day 1)
* 4 weeks after treatment start (day 29)
* 8 or 12 weeks after treatment start and every 8 or 12 weeks thereafter (i.e. at the same time of each imaging tumour assessment) until evidence of progressive disease by RECIST 1.1

For subjects receiving treatments with a 3-weekly schedule, blood and plasma samples for ctDNA testing will be collected at the following timepoints:

Blood :

* Before treatment start (day 1)
* 3 weeks after treatment start (day 22)

Plasma :

* Before treatment start (day 1)
* 6 weeks after treatment start (day 43)
* 8 or 12 weeks after treatment start and every 8 or 12 weeks thereafter (i.e. at the same time of each imaging tumour assessment) until evidence of progressive disease by RECIST 1.1

ctDNA analyses will be done in a centralised laboratory (Foundation Medicine Inc). Full report of the ctDNA analysis will be provided to the study team to allow correlation with clinical data and exploratory analyses. The results of the ctDNA analysis will not be communicated to the treating physician (with the only exception of the analysis by F1CDx on tumour tissue at screening) and therefore will not have any impact on treatment decision (i.e., all study subjects will be treated according to standard practice).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Male or female
3. ECOG performance status ≤2
4. Must have histologically or cytologically verified colorectal cancer adenocarcinoma
5. Inoperable locally advanced or metastatic disease
6. Presence of measurable disease (by RECIST criteria version 1.1) on baseline CT scan of the thorax/abdomen/pelvis or CT scan of the thorax and MRI of the abdomen/pelvis
7. At least two prior systemic treatments for advanced/metastatic colorectal cancer including oxaliplatin and irinotecan-based therapy (adjuvant or neoadjuvant systemic chemotherapy will be considered if tumour progression was documented within 6 month of the last chemotherapy dose)
8. Candidate for standard third-line or subsequent lines of therapy as per decision of the treating physician
9. Life expectancy of at least 3 months
10. Women of childbearing potential must have a negative serum pregnancy test done within 28 days prior to enrolment.
11. Effective contraception is in place for women of childbearing potential.
12. Completion of all necessary screening procedures within 28 days prior to enrolment.
13. Availability of archived tumour tissue
14. Signed Informed Consent form (ICF) obtained prior to any study related procedure.

    Inclusion criterion applicable to FRANCE only
15. Affiliated to the French Social Security System

Exclusion Criteria:

1. Tumours other than colorectal cancer
2. Histologies other than adenocarcinoma
3. Any baseline medical condition that would contraindicate the use of systemic chemotherapy or may preclude the regular administration of the same
4. Any psychiatric condition that would prohibit the understanding or rendering of informed consent
5. Other invasive malignancy within 3 years except for non-invasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured
6. Subject with a significant medical, neuro-psychiatric, or surgical condition, currently uncontrolled by treatment, which, in the principal investigator's opinion, may interfere with completion of the study.
7. Pregnant and/ or lactating women

   Exclusion criterion applicable to FRANCE only
8. Vulnerable persons according to the article L.1121-6 of the Public Health Code, adults who are the subject of a measure of legal protection or unable to express their consent according to article L.1121-8 of the Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-04-12 (Estimated); Study Completion 2026-12-12 (Estimated)

PRIMARY OUTCOMES:
Optimal timepoint and cut-off value for early on-treatment ctDNA changes | at 2 or 3 weeks
  To select the optimal timepoint and cut-off value for early on-treatment ctDNA changes (as assessed by F1Monitor) that predict progressive disease as best radiological response with a high degree of specificity.

SECONDARY OUTCOMES:
optimal timepoint and cut-off value for on-treatment ctDNA changes at 4 or 6 weeks | Day 29 or 43
  To select the optimal timepoint and cut-off value for on-treatment ctDNA changes at 4 or 6 weeks (as assessed by F1Monitor) that predict progressive disease as best radiological response with a high degree of specificity.
rapid turnaround time of ctDNA testing based on F1LCDx | through study completion, an average of 1 year
  To demonstrate rapid turnaround time of ctDNA testing based on F1LCDx and identify technical or logistical challenges to the implementation of an on-treatment ctDNA-driven treatment approach in a follow-on study.
tumour heterogeneity | Day 1
  To evaluate tumour heterogeneity before treatment start as assessed by F1CDx in the tumour tissue and F1LCDx in the whole blood.
CGP changes during treatment | Day 1 and 15 or D1 and D22
  To track CGP changes during treatment as assessed by F1LCDx.

OTHER OUTCOMES:
exploratory genomics and radiomics profiles associated with progresdsive disease as best radiological response | through study completion, an average of 1 year
  To characterize the positive predictive value of baseline genomic and radiomic profiles for tumour progression at the first radiological assessment
prognostic value of ctDNA. | through study completion, an average of 1 year
  To confirm the prognostic value of ctDNA.

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (5):
  - Institut Jules Bordet, Anderlecht
  - UZ Antwerpen, Antwerp
  - CHIREC Delta, Brussels
  - CHU Ambroise Pare, Mons
  - Cliniques Universitaires Saint Luc, Woluwe-Saint-Lambert
- France (7):
  - Centre Georges François Leclerc, Dijon
  - Hopital Franco-Britannique - Fondation Cognacq-Jay, Levallois-Perret
  - Hopital privé Jean Mermoz, Lyon
  - Hopital St-Louis, Paris
  - CHU Poitiers, Poitiers
  - ICO Saint-Herblain, Saint-Herblain
  - ICANS Strasbourg, Strasbourg

REFERENCES:
- [Derived] Assaf I, Bregni G, Anthoine G, Aparicio T, Artru P, Abdelghani MB, Buyse M, Chibaudel B, Coart E, Diaz M, Evrard C, Geboes K, Ghiringhelli F, Puleo F, Raimbourg J, Vandamme T, Van den Eynde M, Hendlisz A, Sclafani F. Rationale and Design of the COPERNIC Trial: A Study of On-treatment ctDNA Changes in Chemo-refractory Colorectal Cancer Patients. Clin Colorectal Cancer. 2025 Mar;24(1):101-105. doi: 10.1016/j.clcc.2024.08.004. Epub 2024 Sep 3. PMID 39341700